CLINICAL TRIAL: NCT01986829
Title: Tumor Ablation in Metastatic Sarcoma Stable on Chemotherapy
Brief Title: Cryoablation, Radiofrequency Ablation, or Microwave Ablation in Treating Patients With Metastatic Sarcoma Stable on Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201309108
Record Dates: First submitted 2013-11-11; First posted 2013-11-19 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Osteosarcoma; Sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (ablation) (Experimental): * Patients undergo cryoablation, radiofrequency ablation, or microwave ablation of each lesion.
  * Patients complete pain survey (BPI-Short form) and quality of life questionnaires (FACT-G7)
  Interventions: Device: Microwave ablation; Device: Cryoablation; Device: Radiofrequency ablation; Other: BPI-Short form; Other: FACT-G7

INTERVENTIONS:
Device: Microwave ablation — * Microwave ablation will be predominantly used on metastatic soft tissue lesions and will include use of Covidien's Evident™ MWA System. Microwave ablation is performed under ultrasound, CT, and occasional fluoroscopic guidance with CT fluoroscopy available for intermittent use in probe placement and CT monitoring of ablation.
  * Microwave antennae from Covidien (Mansfield, MA) are either introduced into the lesion co-axially through a bone biopsy needle or directly into the lesions that are amenable to such, i.e., soft tissue, lung, liver, and large lytic lesions with extensive bone destruction.
Device: Cryoablation — * Cryoablation is performed under ultrasound, CT and occasional fluoroscopic guidance with CT fluoroscopy available for intermittent use in cyroprobe placement and CT monitoring of ablation.
  * Cryoprobes from Endocare Inc. (Irvine CA) or Galil Medical (Arden Hills MN) are either introduced into the lesion co-axially through a bone biopsy needle or directly into the lesions that are amenable to such, i.e., soft tissue, lung, liver, and large lytic lesions with extensive bone destruction.
  Other Names: Cryosurgery; Cryosurgical ablation
Device: Radiofrequency ablation — -Radiofrequency ablation will be predominantly used on metastatic spine lesions and will include use of the Dfine STAR ablation probe. This probe will be placed coaxially through an introducer needle into the spinal metastatic lesion.
Other: BPI-Short form — -Prior to ablation, 1 day post-ablation, 1 month post-ablation (from first procedure if more than 1 is done), and time of disease progression
Other: FACT-G7 — -Prior to ablation, 1 day post-ablation, 1 month post-ablation (from first procedure if more than 1 is done), and time of disease progression

SUMMARY:
This phase II trial studies how well cryoablation, radiofrequency ablation, or microwave ablation works in treating patients with metastatic sarcoma stable on chemotherapy. Cryoablation kills tumor cells by freezing them. Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Microwave ablation kills tumor cells by heating them to several degrees above body temperature.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high-grade metastatic sarcoma that has been stable on 6-12 cycles of one chemotherapeutic regimen (cytotoxic or biologic) although a change in chemotherapy is allowed if it is a result of toxicity/tolerability rather than progression. A patient must not have evidence of progression at any time while on chemotherapy in order to be eligible for this trial.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, PET CT, or MRI exam.
* At least 18 years of age.
* ECOG performance status ≤ 2 (Karnofsky ≥60%)
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN or 3x IULN with normal ALT and AST in patients with Gilbert's disease
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine less than the institutional upper limit of normal OR creatinine clearance ≥ 50 mL/min/1.73 m2
  * INR<1.5 or patient off Coumadin at the time of ablation
* No more than 10 treatable lesions as evaluated by an experienced interventional oncologic radiologist for eligibility and lesion accessibility as the ablation of more than 10 lesions becomes technically infeasible. These lesions must be treated in a two- to three-week time period from initial interventional radiology evaluation. Lung and liver lesions can range from 1 cm to 7 cm for a single lesion and no greater than 5 cm for multiple lesions. There are no size criteria for the osseous lesions.
* The lesions will be amenable to a safe, ultrasound/computed tomographic/fluoroscopic guided percutaneous approach. The targeted metastases must be sufficiently separable from the central nervous system, major peripheral motor nerves, bowel, and bladder. All lesions must be amenable to treatment.
* If patients have received radiation therapy, there must be a one-month washout period.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of ablation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria

* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or localized prostate cancer.
* Receiving any other investigational agents simultaneously or within 3 weeks following ablation procedure.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding.
* Patients whose treatment plans include continuing chemotherapy after ablation as per the treating physician, as ablation therapy is meant to serve as maintenance therapy in lieu of chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Van Tine, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirbe AC, Jennings J, Saad N, Giardina JD, Tao Y, Luo J, Berry S, Toeniskoetter J, Van Tine BA. A Phase II Study of Tumor Ablation in Patients with Metastatic Sarcoma Stable on Chemotherapy. Oncologist. 2018 Jul;23(7):760-e76. doi: 10.1634/theoncologist.2017-0536. Epub 2018 Feb 27. PMID 29487221
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/03/2014 and closed to participant enrollment on 06/19/2017.
Period: Overall Study
Arm/Group | Treatment (Ablation)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ablation)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Rate
Description: Defined as the percentage of patients with no progression (local recurrence of an ablated lesion or the appearance of a new lesion) after ablation.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ablation)
Number analyzed (Participants) | 8
Participants | 6

2. Secondary Outcome: Overall Survival (OS)
Description: -Defined as time from diagnosis of metastatic disease to the time of death
Time Frame: Assessed up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ablation)
Number analyzed (Participants) | 9
months | 23.6 [5.1 to 44.5]

3. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Participant's Lack of Energy
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I have a lack of energy"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: -2 participants were not evaluable for the outcome measures as they did not complete the surveys. An additional participant did not complete the survey at progression. 2 additional participants did not progress and did not complete the surveys at disease progression.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-treatment; Post-Treatment; Disease Progression: * Patients undergo cryoablation, radiofrequency ablation, or microwave ablation of each lesion.
  * Patients complete pain survey (BPI-Short form) and quality of life questionnaires (FACT-G7)
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 0 | 2 | 0
  A little bit (score = 1) | 2 | 1 | 2
  Somewhat (score = 2) | 2 | 3 | 1
  Quite a bit (score = 3) | 1 | 1 | 1
  Very much (score = 4) | 2 | 0 | 0

4. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Participant's Nausea
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I have nausea"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 5 | 6 | 2
  A little bit (score = 1) | 1 | 1 | 0
  Somewhat (score = 2) | 1 | 0 | 1
  Quite a bit (score = 3) | 0 | 0 | 1
  Very much (score = 4) | 0 | 0 | 0

5. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Participant's Worry That the Condition Will Get Worse
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I worry that my condition will get worse"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 3 | 2 | 0
  A little bit (score = 1) | 2 | 4 | 2
  Somewhat (score = 2) | 1 | 0 | 1
  Quite a bit (score = 3) | 0 | 1 | 0
  Very much (score = 4) | 1 | 0 | 1

6. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Ability of the Participant to Enjoy Life
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I am able to enjoy life"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: -2 participants were not evaluable for the outcome measure as they did not complete the surveys. 1 participant did not complete this question on the survey at pre-treatment. An additional participant did not complete the survey at progression. 2 additional participants did not progress and did not complete the surveys at disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 6 | 7 | 4
Participants
  Not at all (score = 0) | 0 | 0 | 0
  A little bit (score = 1) | 0 | 2 | 0
  Somewhat (score = 2) | 3 | 0 | 0
  Quite a bit (score = 3) | 1 | 0 | 2
  Very much (score = 4) | 2 | 5 | 2

7. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Ability of the Participant to Sleep Well
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I am sleeping well"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: -2 participants were not evaluable for the outcome measure as they did not complete the surveys. An additional participant did not complete the survey at progression. 2 additional participants did not progress and did not complete the surveys at disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 0 | 0 | 0
  A little bit (score = 1) | 2 | 2 | 2
  Somewhat (score = 2) | 2 | 3 | 1
  Quite a bit (score = 3) | 1 | 1 | 1
  Very much (score = 4) | 2 | 1 | 0

8. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Contentment of the Participant's Qualify of Life
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I am content with the quality of my life right now"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 0 | 0 | 0
  A little bit (score = 1) | 1 | 0 | 0
  Somewhat (score = 2) | 1 | 0 | 0
  Quite a bit (score = 3) | 5 | 4 | 3
  Very much (score = 4) | 0 | 3 | 1

9. Secondary Outcome: Change in Quality of Life (QOL) Following Ablation Procedure as Measured by the Participant's Pain
Description: * Measured with the FACT-G7 validated survey. Final assessment at time of disease progression.
  * The question participant was asked was "I have pain"
  * 7 questions about quality of life with answers that range from 0=not at all to 4 = very much
  * Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean QOL scores between any two times. All analyses will be two-sided at a significance level of 0.05. This statistical analysis was not able to be performed due to the sample size being too small.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Post-Treatment | Disease Progression
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Not at all (score = 0) | 2 | 2 | 1
  A little bit (score = 1) | 5 | 1 | 3
  Somewhat (score = 2) | 0 | 2 | 0
  Quite a bit (score = 3) | 0 | 0 | 0
  Very much (score = 4) | 0 | 2 | 0

10. Secondary Outcome: Change in Pain Following Ablation Procedure
Description: Measured using the Brief Pain Inventory. Final assessment at time of disease progression. Generalized estimating equation (GEE) analysis will be used to take into account the correlation of repeated measures from the same subject. Contrast statements will be used to compare mean BPI scores between any two times. All analyses will be two-sided at a significance level of 0.05.
Time Frame: Pre-treatment (baseline), post-treatment (1-month post ablation), and disease progression (up to 5 years post-ablation)
Population: The data for this outcome measure was not collected as participant's pain was collected via the Fact G7 questionnaire.
Arm/Group | Treatment (Ablation)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on the first day of ablation through 30 days following the completion of ablation.
Arm/Group | Treatment (Ablation)
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ablation) (N=9)
Intraoperative hemorrhage (Blood and lymphatic system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ablation) (N=9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT01986829/Prot_SAP_000.pdf